CLINICAL TRIAL: NCT03053830
Title: An Open Label Study of the Effects of Ketamine on a Veteran Clinical Population With Major Depressive Disorder (MDD)
Brief Title: Open Label Ketamine Treatment for Major Depressive Disorder in Veterans
Acronym: Ket-MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mohini Ranganathan, MD, MD, VA Connecticut Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR0012
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Group (Experimental): Veterans with Major Depressive Disorder getting up to 6 infusions of 0.5mg/kg ketamine in normal saline; one infusion per week, 40 minutes per infusion with time points lasting up to 5 hours.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 0.5mg/kg ketamine in normal saline. Infusion will be delivered during a 40 minute interval

SUMMARY:
Medically healthy Veterans ages 21-75 that have been diagnosed with Depression will get up to 6 treatments of Ketamine infusions, weekly. After treatment is completed, follow up will occur at 1 month, 3 months, and 6 months after completion of infusions to evaluate the longer term effects of ketamine.

DETAILED DESCRIPTION:
A total of 25 depressed subjects between the ages of 21-75 who have current major depressive disorder without psychotic features by DSM-5 will be recruited. Subjects will be accepted into the protocol after an opportunity to review and provide voluntary written informed consent and completion of a comprehensive medical and psychiatric history, physical examination, mental status examination, and routine laboratory assessments. Patients will be recruited in outpatient settings to the Refractory Depression Clinic. Providers or Refractory Depression consult team will be informed if the patient may be eligible for participation in the ketamine protocol. Subjects must have established care in the VA Connecticut Healthcare System. If the Veteran is interested, a screening visit for further evaluation for the ketamine protocol will be scheduled. Veterans will receive up to 6 infusions for ketamine weekly, per PI discretion. The primary goal of this proposal is to test the effectiveness of repeated ketamine treatment (0.5 mg/kg; once or twice a week for up to 6 weeks; up to a total of 6 ketamine infusions). An open-label trial will be conducted that will include up to 25 Veterans with MDD with a follow-up of 6 months. This open-label trial will allow us to examine the safety and tolerability of the ketamine treatment in this population and the long-term effects. All patients will receive usual standard care during this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 21-75 years old
2. Current major depressive disorder without psychotic features by DSM-5
3. Montgomery-Åsberg Depression Rating Scale (MADRS) ≥ 20
4. Able to provide written informed consent

Exclusion Criteria:

1. Current or past history of psychotic features or psychotic disorder
2. Current or past history of delirium or dementia
3. Current uncontrolled hypertension (systolic BP > 170 mm Hg or diastolic BP > 100 mm Hg)
4. Unstable medical condition or allergy to ketamine or lorazepam---clinically determined by a physician
5. Pregnant or nursing women, positive pregnancy test, or inadequate birth control methods in women of childbearing potential
6. Positive opioid or illicit drug screen test (except marijuana)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, 40 mins after infusion, 140 mins after infusion, 240 mins after infusion
  MADRS is a standardized instrument to ascertain depressed mood and neurovegetative signs and symptoms of a major depressive episode.
Change in Quick Inventory of Depressive Symptomatology-Self Report (QUIDS-SR) | Baseline, 40 mins after infusion, 80 mins after infusion, 110 mins after infusion, 240 mins after infusion
  A patient rated depression instrument
Change in Hamilton Anxiety Rating Scale (HAM-A) | Frame: Baseline, 40 mins after infusion,140 mins after infusion, 240 mins after infusion
  Standardized instrument to evaluate anxiety severity
Clinical Global Impression Scale | Baseline
  Widely used instrument which asses overall severity of illness on a 1-7 point scale, with 1 indicating, not at all ill and 7 indicating among the most extremely ill patients
Change in Brief Psychotic Rating Scale (BPRS) | Baseline, 40 mins after infusion, 80 mins after infusion, 110 mins after infusion, 140 mins after infusion, 240 mins after infusion
  The BPRS is a standardized instrument that contains scales assessing psychotic symptoms including positive and negative symptoms, activation and emotional distress.
Change in Clinician-Administered Dissociative States Scale (CADSS) | Baseline, 40 mins after infusion, 80 mins after infusion, 110 mins after infusion, 140 mins after infusion, 240 mins after infusion
  The CADSS has self and interviewer-administered items including 5 subscales, generated a priori, evaluating dissociation including altered environmental perception, time perception, spatial/body perception, derealization and memory impairment.
Change in Visual Analog Scale (VAS) of Mood States | Baseline, 40 mins after infusion, 80 mins after infusion, 110 mins after infusion, 140 mins after infusion, 240 mins after infusion
  The VAS includes scales for anxiety, drowsiness, high irritability, anger and sadness. The scales are 100 mm lines marked by subjects at a point corresponding to the apparent intensity of the feeling state (0 = none, to 100 = most ever).
Time Line Follow Back (TLFB) | Baseline
  The TLFB is a standardized measure utilized for collecting information on daily alcohol use as well as other substance use.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline
  The C-SSRS has both lifetime/recent and since last visit versions. The "Lifetime/Recent" version gathers information on lifetime history of suicidality and recent suicidal ideation/self-injurious behavior. The "Since Last Visit" version of the C-SSRS asks about any suicidal thoughts or behaviors the subject has exhibited since the last time administered the C-SSRS.
Quality of life enjoyment and satisfaction survey (Q-LES-Q) | Baseline
  The Q-LES-Q is a self-report measure of quality of life.
Cognition | 140 mins after infusion
  A standard computerized battery will be done to assess cognitive ability post treatment of ketamine. The battery will include a wide range on cognitive tasks including but not
  limited to attention, learning, and working memory. While it is know ketamine causes acute cognitive effects, the longer-term effects of ketamine are not known. When the cognitive battery is being conducted on test days it will be done at the end of the test day, to eliminate the confounding effects of acute treatment of ketamine..

CONTACTS AND LOCATIONS:
Locations (1):
- VA Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.